CLINICAL TRIAL: NCT01729806
Title: A Phase I Study of Ipilimumab in Combination With Rituximab in Patients With Relapsed/Refractory CD20+ B-Cell Lymphoma
Brief Title: Ipilimumab and Rituximab in Treating Patients With Relapsed or Refractory B-cell Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02213; NCI-2012-02213 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); PHI-69; CDR0000743246; NCI# 9197; 9197 (Other: City of Hope Comprehensive Cancer Center); 9197 (Other: CTEP); P30CA033572 (NIH); U01CA062505 (NIH); UM1CA186704 (NIH); UM1CA186717 (NIH)
Record Dates: First submitted 2012-11-14; First posted 2012-11-20 (Estimated); Last update posted 2018-04-11 (Actual); Status verified 2018-04

CONDITIONS: CD20 Positive; Recurrent B-Cell Non-Hodgkin Lymphoma; Refractory B-Cell Non-Hodgkin Lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell | interventions — Ipilimumab; CTLA-4 Antigen; Rituximab; CT-P10

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A (ipilimumab and rituximab) (Experimental): Patients receive rituximab IV over 2-6 hours once weekly in weeks 1-4 and ipilimumab IV over 90 minutes once weekly in weeks 1, 4, 7, and 10. Patients then receive ipilimumab IV over 90 minutes and rituximab IV over 2-6 hours once every 12 weeks for up to 1 year in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Ipilimumab; Other: Laboratory Biomarker Analysis; Biological: Rituximab
- Arm B (ipilimumab and rituximab) (Experimental): Patients receive rituximab IV over 2-6 hours once weekly in weeks 1-4 and ipilimumab IV over 90 minutes once weekly in weeks 3, 6, 9, and 12. Patients then receive ipilimumab IV over 90 minutes and rituximab IV over 2-6 hours once every 12 weeks for up to 1 year in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Ipilimumab; Other: Laboratory Biomarker Analysis; Biological: Rituximab

INTERVENTIONS:
Biological: Ipilimumab — Given IV
  Other Names: Anti-Cytotoxic T-Lymphocyte-Associated Antigen-4 Monoclonal Antibody; BMS-734016; MDX-010; MDX-CTLA4; Yervoy
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: Rituximab — Given IV
  Other Names: ABP 798; BI 695500; C2B8 Monoclonal Antibody; Chimeric Anti-CD20 Antibody; CT-P10; IDEC-102; IDEC-C2B8; IDEC-C2B8 Monoclonal Antibody; MabThera; Monoclonal Antibody IDEC-C2B8; PF-05280586; Rituxan; Rituximab Biosimilar ABP 798; Rituximab Biosimilar BI 695500; Rituximab Biosimilar CT-P10; Rituximab Biosimilar GB241; Rituximab Biosimilar IBI301; Rituximab Biosimilar PF-05280586; Rituximab Biosimilar RTXM83; Rituximab Biosimilar SAIT101; RTXM83

SUMMARY:
This partially randomized phase I trial studies the side effects and best dose of ipilimumab when given together with rituximab in treating patients with B-cell lymphoma that has returned or has not responded to treatment. Monoclonal antibodies, such as ipilimumab and rituximab, may interfere with the ability of cancer cells to grow and spread.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine a recommended phase II dose for ipilimumab in combination with rituximab.

SECONDARY OBJECTIVES:

I. To obtain preliminary information on the effect of adding ipilimumab to rituximab in regard to: immune response; clinical anti-tumor response/overall remission rate (ORR) (complete remission + partial remission); progression free survival (PFS).

OUTLINE: This is a dose-escalation study of ipilimumab followed by a randomized study.

PART I:

INDUCTION: Patients receive ipilimumab intravenously (IV) over 90 minutes once every 3 weeks for 12 weeks and rituximab IV over 2-6 hours once weekly for 4 weeks.

MAINTENANCE: Patients receive ipilimumab IV over 90 minutes and rituximab IV over 2-6 hours once every 12 weeks for up to 1 year.

PART II: Patients are randomized to 1 of 2 treatment arms.

ARM A: Patients receive rituximab IV over 2-6 hours once weekly in weeks 1-4 and ipilimumab IV over 90 minutes once weekly in weeks 1, 4, 7, and 10. Patients then receive ipilimumab IV over 90 minutes and rituximab IV over 2-6 hours once every 12 weeks for up to 1 year in the absence of disease progression or unacceptable toxicity.

ARM B: Patients receive rituximab IV over 2-6 hours once weekly in weeks 1-4 and ipilimumab IV over 90 minutes once weekly in weeks 3, 6, 9, and 12. Patients then receive ipilimumab IV over 90 minutes and rituximab IV over 2-6 hours once every 12 weeks for up to 1 year in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Previously treated, histologically confirmed cluster of differentiation (CD)20+ B cell lymphoma; bone marrow biopsies as the sole means of diagnosis are not acceptable, but they may be submitted in conjunction with nodal biopsies or extra nodal biopsies; fine needle aspirates are not acceptable
* All patients must be informed of the investigative nature of the clinical trial and give written informed consent in accordance with institutional and federal guidelines
* Able to adhere to the study visit schedule and other protocol requirements
* Karnofsky >= 70%
* Life expectancy expected to be greater than 3 months
* Leukocytes >= 3,000/mcL
* Absolute neutrophil count >= 1,000/mcL
* Platelets >= 50,000/mcL
* Total bilirubin =< 2.0 x institutional upper limit of normal
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x institutional upper limit of normal
* Serum creatinine =< 2.0 x upper limit of normal OR calculated creatinine clearance >= 30 ml/min/1.73 M^2 by the modified Cockcroft and Gault formula OR creatinine clearance >= 30 mL/min obtained from a 24-hour urine collection
* At least one measurable lesion according to international workshop lymphoma response criteria; there must be measurable lymphadenopathy to follow with serial exam and/or imaging
* All previous cancer therapy, including radiation, hormonal therapy and surgery, must have been discontinued at least 4 weeks prior to treatment in this study
* Patients must have evidence of progression of disease during or after last treatment
* Submission of original biopsy for review and verification by participating center hematopathologist
* Disease free of prior malignancies for >= 3 years with exception of currently treated basal cell, squamous cell carcinoma of the skin, or carcinoma "in situ" of the cervix or breast

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier
* Patients with a history of prior treatment with ipilimumab
* Patients with a history of prior treatment with an anti-programmed cell death (PD) 1 antibody, CD137 agonist or other immune activating therapy such as anti-CD 40 antibody are excluded unless 5 half-lives of the agent (minimum of 8 weeks) have intervened since the therapy; patients who have received prior vaccine therapy are eligible
* Patients who are receiving any other investigational agents
* Autoimmune disease: patients with a history of inflammatory bowel disease, including ulcerative colitis and Crohn's disease, are excluded from this study, as are patients with a history of symptomatic disease (e.g., rheumatoid arthritis, systemic progressive sclerosis [scleroderma], systemic lupus erythematosus, autoimmune vasculitis [e.g., Wegener's granulomatosis]); central nervous system (CNS) or motor neuropathy considered of autoimmune origin (e.g. Guillain-Barre syndrome and myasthenia gravis, multiple sclerosis)
* Patients with known immune impairment who may be unable to respond to anti-cytotoxic T-lymphocyte antigen 4 (CTLA 4) antibody
* Patients with known uncontrolled brain metastases are excluded; however, patients with stable brain disease (off corticosteroids) at least 2 weeks after completion of appropriate therapy for their brain metastases are eligible
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to rituximab
* Patients on systemic corticosteroids (except for patients on stable doses of hormone replacement therapy such as hydrocortisone), or other immunosuppressants (e.g., infliximab, mycophenolate mofetil) are excluded
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Patients with chronic human immunodeficiency virus (HIV), hepatitis B or hepatitis C infections are excluded
* Pregnant women are excluded from this study
* HIV-positive patients on combination antiretroviral therapy are ineligible
* Rituximab within six weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2012-11-19 (Actual); Primary Completion 2018-03-30 (Actual); Study Completion 2018-03-30 (Actual)

PRIMARY OUTCOMES:
Incidence of toxicities according to the Common Terminology Criteria for Adverse Events version 4 | Up to 12 months
  Tables will be created to summarize the toxicities and side effects by dose, course, organ and severity.

SECONDARY OUTCOMES:
Immune response as measured by the frequency of activated T-cells, absolute lymphocyte count, antibody dependent cell-mediated cytotoxicity, and kinetics and magnitude of B-cell depletion | Up to 14 weeks
  Regression methods (adapted for repeated measures) will be used to describe the changes over time. In addition to summarizing the changes over time within each arm, these regression models will contain contrasts to compare the two arms in terms of changes.
Clinical anti-tumor response (complete response and partial response as per international workshop lymphoma response criteria [Cheson 2007]) | Up to 12 months
Progression-free survival | From when the patient started treatment to the time the patient is first recorded as having disease relapse/progression, or to the date of death if the patient dies due to causes other than disease progression, assessed up to 12 months
  Progression-free survival will be summarized using Kaplan-Meier plots.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Tuscano, Principal Investigator — City of Hope Comprehensive Cancer Center
Locations (7):
- United States (7):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - City of Hope South Pasadena, South Pasadena, California
  - Washington University School of Medicine, St Louis, Missouri
  - Duke University Medical Center, Durham, North Carolina
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania